CLINICAL TRIAL: NCT04707768
Title: A Randomized, Open-label, Active-controlled Study Evaluating the Efficacy and Safety of Dose Conversion From a Long-acting Erythropoiesis-stimulating Agent (Mircera®) to Three Times Weekly Oral Vadadustat for the Maintenance Treatment of Anemia in Hemodialysis Subjects
Brief Title: Study Evaluating the Efficacy and Safety of Dose Conversion From a Long-acting Erythropoiesis-stimulating Agent (Mircera®) to Three Times Weekly Oral Vadadustat for the Maintenance Treatment of Anemia in Hemodialysis Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AKB-6548-CI-0039
Record Dates: First submitted 2021-01-12; First posted 2021-01-13 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Anemia Associated With Chronic Kidney Disease (CKD)
Keywords: Anemia; Chronic Kidney Disease; CKD; Hemodialysis; Vadadustat; Erythropoiesis-stimulating agent (ESA)
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — vadadustat; continuous erythropoietin receptor activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vadadustat low dose (Experimental): Participants previously receiving Mircera® received vadadustat for up to 52 weeks with an initial dose of 600 milligrams (mg).
  Interventions: Drug: Vadadustat
- Vadadustat high dose (Experimental): Participants previously receiving Mircera® received vadadustat for up to 52 weeks with an initial dose of 900 mg.
  Interventions: Drug: Vadadustat
- Mircera® (Active Comparator): Participants will continue to receive Mircera® for up to 52 weeks.
  Interventions: Drug: Mircera®

INTERVENTIONS:
Drug: Vadadustat — oral tablets
  Arms: Vadadustat high dose; Vadadustat low dose
Drug: Mircera® — intravenous administration
  Arms: Mircera®

SUMMARY:
This study will be conducted to demonstrate the efficacy and safety of vadadustat administered three times weekly (TIW) compared to a long-acting erythropoiesis-stimulating agent (ESA) (Mircera®) for the maintenance treatment of anemia in hemodialysis participants.

DETAILED DESCRIPTION:
Following randomization, there will be 2 periods during the study:

* Conversion and Maintenance Period (Weeks 0 to 52): There will be a primary efficacy evaluation period (Weeks 20 to 26) and a secondary efficacy evaluation period (Weeks 46 to 52).
* Safety Follow-up Period (Early Termination [ET] and Follow-Up): post-treatment safety follow-up visit (ET/End of Treatment [EOT] +4 weeks) either in person or via telephone.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Receiving chronic, outpatient in-center hemodialysis three times weekly (TIW) for end-stage kidney disease for at least 12 weeks prior to Screening Visit 1 (SV1)
* Currently maintained on Mircera® (≤250 μg/month) with at least 2 doses received within 8 weeks prior to Screening Visit 2 (SV2)
* Mean Screening hemoglobin (Hb) between 8.5 and 11.0 grams per deciliter (g/dL) (inclusive), as determined by the average of 2 Hb values measured by the central laboratory at least 4 days apart between SV1 and SV2
* Serum ferritin ≥100 nanograms per milliliter (ng/mL) and transferrin saturation (TSAT) ≥20% during Screening
* Folate and vitamin B12 measurements ≥ lower limit of normal during Screening

Exclusion Criteria:

* Anemia due to a cause other than chronic kidney disease (CKD).
* Clinically meaningful bleeding event within 8 weeks prior to Baseline
* Red blood cell (RBC) transfusion within 8 weeks prior to Baseline
* Having received any doses of darbepoetin alfa (Aranesp®) within 4 weeks prior to Baseline
* Having received any doses of epoetin alfa (Epogen®) within 1 week prior to Baseline.
* Current uncontrolled hypertension.
* Acute coronary syndrome (hospitalization for unstable angina or myocardial infarction), surgical or percutaneous intervention for coronary, cerebrovascular or peripheral artery disease (aortic or lower extremity), surgical or percutaneous valvular replacement or repair, sustained ventricular tachycardia, hospitalization for heart failure (HF) or New York Heart Association Class IV HF, or stroke within 12 weeks prior to or during Screening.
* Known hypersensitivity to vadadustat, Mircera®, or any of their excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Akebia Therapeutics Inc.
Locations (55):
- United States (55):
  - Research Site, Huntsville, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Pine Bluff, Arkansas
  - Research Site, El Centro, California
  - Research Site, Escondido, California
  - Research Site, Fresno, California
  - Research Site, Granada Hills, California
  - Research Site, Porterville, California
  - Research Site, San Diego, California
  - Research Site, Arvada, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Hockessin, Delaware
  - Research Site, Bradenton, Florida
  - Research Site, Coral Gables, Florida
  - Research Site#1, Coral Springs, Florida
  - Research Site#2, Coral Springs, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Athens, Georgia
  - Research Site, Buford, Georgia
  - Research Site, Dalton, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Nampa, Idaho
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Plymouth, Massachusetts
  - Research Site, Springfield, Massachusetts
  - Research Site, Kalamazoo, Michigan
  - Research Site, Rochester Hills, Michigan
  - Research Site, Saint Clair Shores, Michigan
  - Research Site, Brookhaven, Mississippi
  - Research Site, Columbus, Mississippi
  - Research Site, Tupelo, Mississippi
  - Research Site, North Platte, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Portsmouth, New Hampshire
  - Research Site, Albuquerque, New Mexico
  - Research Site, Gallup, New Mexico
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Kinston, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Kittanning, Pennsylvania
  - Research Site, Knoxville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Mansfield, Texas
  - Research Site, Mission, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Alexandria, Virginia
  - Research Site, Salem, Virginia
  - Research Site, Woodbridge, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toka HR, Bernardo M, Burke SK, Luo W, Manllo-Karim R, Ullah I, Yang Z, Zhang Z, Tumlin J. Vadadustat Three Times Weekly in Patients With Anemia Due to Dialysis-Dependent CKD. Am J Kidney Dis. 2025 Apr;85(4):454-464.e1. doi: 10.1053/j.ajkd.2024.09.006. Epub 2024 Nov 7. PMID 39521398
- [Derived] Kooienga L, Burke S, Kathresal A, Luo W, Yang Z, Zhang Z, Zwiech R, Hernandez GT. Safety and Efficacy of Vadadustat Once Daily and Three Times Weekly in Patients With Dialysis-Dependent CKD With Anemia. Kidney360. 2024 Nov 1;5(11):1652-1661. doi: 10.34067/KID.0000000567. Epub 2024 Sep 4. PMID 39231617

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomzied, open-label, active-controlled study of the efficacy and safety of conversion from long-acting Erythropoiesis-stimulating Agent (ESA) (Methoxy polyethylene glycol-epoetin beta [Mircera®]) to vadadustat Three Times Weekly (TIW) for the maintenance treatment of anemia in hemodialysis participants.
Pre-assignment Details: A total of 456 participants were enrolled in the study. Participants were randomized 1:1:1 to Vadadustat 600 milligrams (mg) TIW Vadadustat 900 mg TIW or to remain on Mircera® according to the dialysis center's protocol.
Groups:
- Vadadustat 600 mg TIW: Participants were randomized to receive Vadadustat at an initial oral dose of 600 mg TIW. Up-and-down titration was allowed during the study based on hemoglobin (Hb) level measurements to maintain target Hb level
- Vadadustat 900 mg TIW: Participants were randomized to receive Vadadustat at an initial oral dose of 900 mg TIW. Up-and-down titration was allowed during the study based on Hb level measurements to maintain target Hb level
- Mircera®: Participants were randomized to Mircera® were already on Mircera®, the initial dosing regimen in the study was based on the prior dosing regimen
Period: Overall Study
Arm/Group | Vadadustat 600 mg TIW | Vadadustat 900 mg TIW | Mircera®
Started | 152 | 152 | 152
Completed | 99 | 98 | 118
Not Completed | 53 | 54 | 34
Not completed — Adverse Event | 9 | 18 | 3
Not completed — Investigator's Discretion | 8 | 4 | 3
Not completed — Withdrawal by Subject | 6 | 8 | 2
Not completed — Lack of Efficacy | 1 | 3 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3
Not completed — Death | 13 | 11 | 13
Not completed — Protocol Violation | 2 | 1 | 0
Not completed — Non Compliance with Study Drug | 1 | 0 | 0
Not completed — Transplant | 4 | 4 | 8
Not completed — Other | 9 | 5 | 2

BASELINE CHARACTERISTICS:
Population: Randomized population included all randomized participants.
Groups:
- Vadadustat 600 mg TIW: Participants were randomized to receive Vadadustat at an initial oral dose of 600 mg TIW. Up-and-down titration was allowed during the study based on Hb level measurements to maintain target Hb level
- Total: Total of all reporting groups
Arm/Group | Vadadustat 600 mg TIW | Vadadustat 900 mg TIW | Mircera® | Total
Number analyzed (Participants) | 152 | 152 | 152 | 456
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.4 (14.20) | 61.9 (13.27) | 61.6 (12.80) | 61.0 (13.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 60 | 66 | 194
  Male | 84 | 92 | 86 | 262
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 40 | 56 | 138
  Not Hispanic or Latino | 110 | 109 | 95 | 314
  Unknown or Not Reported | 0 | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 3 | 4 | 12
  Asian | 3 | 2 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 56 | 59 | 53 | 168
  White | 86 | 87 | 92 | 265
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin (Hb) to the Average Over the Primary Evaluation Period (PEP) (Weeks 20 to 26)
Description: The Baseline Hb was defined as the average of last 2 central laboratory Hb measurements of samples taken at or prior to the first dose. The average for the PEP was calculated as the average of all Hb measurements from the central laboratory within the three visit windows during Weeks 20 through 26. Analysis was conducted using an analysis of covariance (ANCOVA) model with multiple imputation for missing data with randomization stratification factors and Baseline Hb as covariates. Change from Baseline was calculated as PEP value minus the Baseline value.
Time Frame: Baseline; Weeks 20 to 26
Population: Randomized Population
Measure: Least Squares Mean (Standard Error); unit: Grams per deciliter (g/dL)
Arm/Group | Vadadustat 600 mg TIW | Vadadustat 900 mg TIW | Mircera®
Number analyzed (Participants) | 152 | 152 | 152
Grams per deciliter (g/dL) | -0.07 (0.095) | 0.14 (0.095) | 0.36 (0.092)

2. Secondary Outcome: Change From Baseline in Hb to the Average Over the Secondary Evaluation Period (SEP) (Weeks 46 to 52)
Description: The Baseline Hb was defined as the average of the last 2 central laboratory Hb values taken on or prior to the first dose date. The average for the SEP was calculated as the average of all Hb measurements from the central laboratory within the three visit windows during Weeks 46 through 52. Analysis was conducted using an ANCOVA model with multiple imputation for missing data with randomization stratification factors and Baseline Hb as covariates. Change from Baseline was calculated as SEP value minus the Baseline value.
Time Frame: Baseline; Weeks 46 to 52
Population: Randomized population.
Measure: Least Squares Mean (Standard Error); unit: Grams per deciliter
Arm/Group | Vadadustat 600 mg TIW | Vadadustat 900 mg TIW | Mircera®
Number analyzed (Participants) | 152 | 152 | 152
Grams per deciliter | -0.11 (0.110) | -0.22 (0.123) | 0.16 (0.102)

ADVERSE EVENTS:
Time Frame: Day 1 through Week 56
Description: Safety Population included all participants who received at least 1 dose of study medication
Arm/Group | Vadadustat 600 mg TIW | Vadadustat 900 mg TIW | Mircera®
All-Cause Mortality (participants affected / at risk) | 14/151 | 12/150 | 17/150
Serious Adverse Events (participants affected / at risk) | 68/151 | 66/150 | 67/150
Other Adverse Events (participants affected / at risk) | 61/151 | 67/150 | 64/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vadadustat 600 mg TIW (N=151) | Vadadustat 900 mg TIW (N=150) | Mircera® (N=150)
COVID 19 (Infections and infestations) | 3 | 5 | 6
COVID 19 pneumonia (Infections and infestations) | 1 | 4 | 8
Pneumonia (Infections and infestations) | 4 | 7 | 2
Sepsis (Infections and infestations) | 2 | 4 | 2
Cellulitis (Infections and infestations) | 1 | 3 | 2
Gangrene (Infections and infestations) | 3 | 0 | 3
Septic shock (Infections and infestations) | 3 | 2 | 1
Osteomyelitis (Infections and infestations) | 4 | 0 | 1
Arteriovenous fistula site infection (Infections and infestations) | 0 | 1 | 2
Bacteraemia (Infections and infestations) | 3 | 0 | 0
Device related sepsis (Infections and infestations) | 0 | 0 | 3
Staphylococcal bacteraemia (Infections and infestations) | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 2
Arteriovenous graft site infection (Infections and infestations) | 0 | 1 | 1
Cellulitis staphylococcal (Infections and infestations) | 0 | 0 | 2
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 1
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 1
Appendiceal abscess (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 0
Asymptomatic COVID 19 (Infections and infestations) | 1 | 0 | 0
Cellulitis gangrenous (Infections and infestations) | 1 | 0 | 0
Chest wall abscess (Infections and infestations) | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis Escherichia coli (Infections and infestations) | 0 | 1 | 0
Herpes zoster meningoencephalitis (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Pancreatic abscess (Infections and infestations) | 0 | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 1 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Varicella zoster virus infection (Infections and infestations) | 0 | 1 | 0
Vascular access site cellulitis (Infections and infestations) | 0 | 1 | 0
Viral sepsis (Infections and infestations) | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 2 | 3 | 11
Acute myocardial infarction (Cardiac disorders) | 4 | 3 | 5
Atrial fibrillation (Cardiac disorders) | 3 | 3 | 3
Cardiac failure congestive (Cardiac disorders) | 5 | 2 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 2 | 1
Cardio respiratory arrest (Cardiac disorders) | 1 | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 2
Pericardial effusion (Cardiac disorders) | 1 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 7 | 6 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 4 | 5
Failure to thrive (Metabolism and nutrition disorders) | 2 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 1 | 3 | 5
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 3 | 2
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 2 | 1
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arteriovenous graft site stenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Haematuria traumatic (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Unintentional medical device removal (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular access malfunction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular graft complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 5
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 4 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 2 | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal polyp (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Mallory Weiss syndrome (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Rectal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 3 | 3
Hypertension (Vascular disorders) | 1 | 1 | 2
Hypertensive emergency (Vascular disorders) | 1 | 1 | 1
Hypertensive urgency (Vascular disorders) | 1 | 1 | 1
Aortic stenosis (Vascular disorders) | 1 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 1 | 0
Shock (Vascular disorders) | 2 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Dry gangrene (Vascular disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 2 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 2
Thalamic infarction (Nervous system disorders) | 0 | 1 | 1
Brain injury (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Hypoxic ischaemic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Seizure like phenomena (Nervous system disorders) | 0 | 0 | 1
Thrombotic stroke (Nervous system disorders) | 0 | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Unresponsive to stimuli (Nervous system disorders) | 1 | 0 | 0
Catheter site thrombosis (General disorders) | 0 | 2 | 0
Death (General disorders) | 0 | 1 | 1
Non cardiac chest pain (General disorders) | 1 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0
Hypothermia (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 3 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0 | 0
Troponin increased (Investigations) | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Benign uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Nephropathy (Renal and urinary disorders) | 0 | 1 | 0
Renal mass (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 2
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Hyperparathyroidism secondary (Endocrine disorders) | 0 | 0 | 1
Blindness transient (Eye disorders) | 1 | 0 | 0
Thrombosis in device (Product Issues) | 0 | 1 | 0
Social stay hospitalisation (Social circumstances) | 0 | 1 | 0
Hospitalisation (Surgical and medical procedures) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vadadustat 600 mg TIW (N=151) | Vadadustat 900 mg TIW (N=150) | Mircera® (N=150)
COVID 19 (Infections and infestations) | 19 | 18 | 19
Diarrhoea (Gastrointestinal disorders) | 16 | 21 | 11
Nausea (Gastrointestinal disorders) | 12 | 13 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 13 | 12
Fall (Injury, poisoning and procedural complications) | 11 | 8 | 11
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 7 | 8 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 8 | 4
Hypertension (Vascular disorders) | 5 | 4 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 5 | 5
Headache (Nervous system disorders) | 3 | 10 | 5
Vomiting (Gastrointestinal disorders) | 4 | 5 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/68/NCT04707768/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/68/NCT04707768/SAP_001.pdf